CLINICAL TRIAL: NCT01097668
Title: SAFETY AND PROOF OF PRINCIPLE STUDY OF ATX-MS-1467 IN PATIENTS WITH RELAPSING MULTIPLE SCLEROSIS: OPEN LABEL UPWARD TITRATION OVER FIVE DOSE LEVELS AND USING TWO ROUTES OF ADMINISTRATION (INTRADERMAL AND SUBCUTANEOUS).
Brief Title: ATX-MS-1467 in Patients With Relapsing Forms of Multiple Sclerosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Apitope Technology (Bristol) Ltd. (Industry)
Collaborators: Aptiv Solutions (Industry); ClinStar, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATX-MS-1467-002
Record Dates: First submitted 2010-03-31; First posted 2010-04-02 (Estimated); Results first posted 2015-02-16 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: Multiple sclerosis; Immunomodulation; Phase 1
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — ATX-MS-1467

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intradermal injection (Experimental): Injections will be given by the intradermal route
  Interventions: Biological: ATX-MS-1467
- Subcutaneous injection (Experimental): Injections will be given by the subcutaneous route
  Interventions: Biological: ATX-MS-1467

INTERVENTIONS:
Biological: ATX-MS-1467 — Disease specific immune modulating treatment for multiple sclerosis

SUMMARY:
Phase 1 study to assess the safety and biological activity of ATX-MS-1467 in patients with relapsing forms of multiple sclerosis. This will be an open label upward dose titration involving injections on 9 occasions, each two weeks apart. After dosing is complete there will be a 22 week follow up period. Blood samples will be drawn throughout the study to monitor safety and the body's response to the injections and MRI scans will be performed on several occasions to follow the course of the multiple sclerosis during the trial.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients who have definite relapsing multiple sclerosis disease as defined by the McDonald criteria (McDonald et al., 2001 and 2005) and as assessed by a neurologist.

  2. HLA DRB1*15 positive.

  3. High baseline levels of T-cell proliferation in response to myelin basic protein, defined as >1000 cpm with a >3 stimulation index compared to background.

  4. Disease duration equal to or less than 10 years (from the first clinical event).

  5. At least one documented relapse in the previous 12 months or two relapses within the previous 24 months prior to screening.

  6. Must be in a clinically stable or improving neurological state during the 28 days preceding Screening.

  7. EDSS score < 5.5.

Exclusion Criteria:

* 1. Subjects treated with β-interferon, plasma exchange, intravenous gamma globulin within the 3 months prior to Study Day 1 2. Subjects treated with glatiramer acetate at any time in the past 3. Subjects who have been treated with parenteral steroids or adrenocorticotropic hormone within 3 months days prior to Study Day 1 4. Prior treatment with: cytotoxic agents (including but not limited to cladribine, mitoxantrone, cyclophosphamide, azathioprine, methotrexate), fingolimod, laquinimod, teriflunomide, total lymphoid irradiation, stem cell or bone marrow transplantation, or monoclonal antibody therapy (including natalizumab, daclizumab, alemtuzumab) 5. Prior use of disease related T-cell vaccine or peptide-tolerising agent to treat MS 6. Use of any investigational drug or experimental procedure within 6 months prior to Study Day 1 including cytokine or anti-cytokine therapy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2010-03; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Chataway, Principal Investigator — National Hospital for Neurology and Neurosurgery, London
Locations (16):
- Russia (11):
  - Municipal Healthcare Institution "City Clinical Hospital #3", Department of neurology, Chelyabinsk
  - State Medical Institution "Republican Clinical Hospital of rehabilitation treatment of Ministry of Healthcare of Tatarstan Republic", Republican clinicodiagnostic center of demyelinating diseases of Ministry of Healthcare of Tatarstan Republic, Kazan'
  - State Educational Institution of Higher Professional Education "1st Moscow State Medical University n.a. I.M. Sechenov of Ministry of Healthcare and Social Development of the Russian Federation, Department of new drugs research, Moscow
  - State Healthcare Institution 'Rostov Regional Clinical Hospital' Center of Neurology, Rostov-on-Don
  - LLC "International Clinic MEDEM", Department of functional diagnostics, Saint Petersburg
  - St. Petersburg State Healthcare Institution "City multifield hospital #2", Department of neurology #2, Saint Petersburg
  - State Educational Institution of Higher Professional Education "St. Petersburg State Medical University n.a. I.V. Pavlov of Roszdrav", Department of neurology with clinic, Saint Petersburg
  - Institution of the Russian Academy of Science "Institute of Human Brain of RAS", Neuroimmunology Laboratory, Saint Petersburg
  - State Healthcare Institution "Samara Regional Clinical Hospital n.a. M.I. Kalinin", Department of neurosurgery, Samara
  - State Educational Institution of Higher Professional Education Saratov State Medical University, Saratov
  - State Educational Institution of Higher Professional Education "Smolensk State Medical Academy of Roszdrav", Department of neurology and neurosurgery based at State Healthcare Institution "Smolensk Regional Clinical Hospital", Smolensk
- United Kingdom (5):
  - North Staffordshire Royal Infirmary, Stoke-on-Trent, Staffordshire
  - National Hospital for Neurology & Neurosurgery, London
  - Queen's Medical Centre, Nottingham
  - Peninsula Medical School, Plymouth
  - Royal Hallamshire Hospital, Sheffield

REFERENCES:
- See also: sponsor — http://www.apitope.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Screening and study procedures were performed at hospital clinics within the United Kingdom and Russian Federation.
Pre-assignment Details: Subjects were human lymphocyte antigen (HLA)-DRB1*15 positive with relapsing-remitting multiple sclerosis as defined by the McDonald criteria and as assessed by a neurologist.
Groups:
- Intradermal Injection; Subcutaneous Injection: Upward titration over 4 dose levels (injections of 25, 50, 100 and 400 ug) of ATX MS 1467 followed by injections of 800 ug injected on 5 occasions. All injections were administered at intervals of 14±3 days.
Period: Overall Study
Arm/Group | Intradermal Injection | Subcutaneous Injection
Started | 21 | 22
Week 20 | 21 (Patient evaluability time point = week 20) | 22 (Patient evaluability time point = week 20)
Week 48 | 19 | 20
Completed | 19 | 20
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: >=18 and <=55 years Gender, female and male
Groups:
- Intradermal Injection: Injections of ATX-MS-1467 given by the intradermal route
- Subcutaneous Injection: Injections of ATX-MS-1467 given by the subcutaneous route
- Total: Total of all reporting groups
Arm/Group | Intradermal Injection | Subcutaneous Injection | Total
Number analyzed (Participants) | 21 | 22 | 43
Age, Continuous [Mean (Full Range); unit: years] | 33.0 [22 to 53] | 31.6 [18 to 52] | 32.3 [18 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 13 | 30
  Male | 4 | 9 | 13
Region of Enrollment [Number; unit: participants]
  Russian Federation | 14 | 20 | 34
  United Kingdom | 7 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability
Description: Occurrence of treatment emergent Adverse Events (AE), Serious Adverse Events, and laboratory abnormalities up to week 48 compared to baseline.
Time Frame: 48 weeks
Population: The Safety population will be denoted as the 'ITT population' for the summarisation of safety endpoints.
Measure: Number; unit: participants
Groups:
- Intradermal Injection: Injections of ATX-MS-1467 administered by the intradermal route
- Subcutaneous Injection: Injections of ATX-MS-1467 administered by the subcutaneous route
Arm/Group | Intradermal Injection | Subcutaneous Injection
Number analyzed (Participants) | 21 | 22
participants | 21 | 22

2. Secondary Outcome: The Effect of ATX-MS-1467 on Brain Magnetic Resonance Imaging (MRI).
Description: Number of new or persisting Gadolinium-enhancing lesions at week 16 and 20 when compared to baseline.
Time Frame: 16 and 20 weeks
Population: ITT population at week 16 and 20 n=21 (Intradermal injection) ITT population at week 16 and 20 n=22 (Subcutaneous injection) MRI population at week 16 and 20 n=17 (Intradermal injection) MRI population at week 16 and 20 n=20 (Subcutaneous injection)
Measure: Mean (95% Confidence Interval); unit: MRI lesions
Groups:
- Intradermal: Injections of ATX-MS-1467 administered by intradermal route
- Subcutaneous Injection: Injections of ATX-MS-1467 administered by subcutaneous route
Arm/Group | Intradermal | Subcutaneous Injection
Number analyzed (Participants) | 21 | 22
MRI lesions
  ITT poulation at baseline | 5.05 [1.83 to 13.93] | 2.09 [0.76 to 5.78]
  ITT population at Week 16 | 0.74 [0.33 to 1.69] | 1.85 [1.00 to 3.41]
  ITT population at Week 20 | 1.65 [0.63 to 4.34] | 1.47 [0.85 to 2.54]
  MRI population at baseline | 3.41 [1.08 to 10.75] | 2.3 [0.79 to 6.71]
  MRI population at Week 16 | 0.73 [0.28 to 1.89] | 1.71 [0.93 to 3.14]
  MRI population at Week 20 | 1.51 [0.48 to 4.73] | 1.20 [0.68 to 2.14]
Statistical Analysis 1: Comparison: Intradermal; Comparison of the baseline 'ITT population' MRI data with week 16 data; Test type: Superiority or Other; p < 0.001, negative binomial model
Statistical Analysis 2: Comparison: Intradermal; Comparison of the baseline 'MRI population' data with data from week 16; Test type: Superiority or Other; p = 0.030, negative binomial model

ADVERSE EVENTS:
Time Frame: Adverse event data collected over the course of the study = 52 weeks
Description: Adverse Events were recorded in the Case Report Form and characterised by severity, relationship to IMP,outcome, action taken, onset and resolution date and seriousness. Occurrences of Multiple Sclerosis relapses were recorded as Adverse Events.
Groups:
- Intradermal Injection - Treatment Emergent: Injections will be administered by the intradermal route
- Subcutaneous Injection - Treatment Emergent: Injections will be administered by the subcutaneous route
- Intradermal Injection - Non Treatment Emergent; Subcutaneous Injection - Non Treatment Emergent: Follow-up period
Arm/Group | Intradermal Injection - Treatment Emergent | Subcutaneous Injection - Treatment Emergent | Intradermal Injection - Non Treatment Emergent | Subcutaneous Injection - Non Treatment Emergent
Serious Adverse Events (participants affected / at risk) | 1/21 | 0/22 | 2/21 | 1/22
Other Adverse Events (participants affected / at risk) | 17/21 | 16/22 | 7/21 | 5/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intradermal Injection - Treatment Emergent (N=21) | Subcutaneous Injection - Treatment Emergent (N=22) | Intradermal Injection - Non Treatment Emergent (N=21) | Subcutaneous Injection - Non Treatment Emergent (N=22)
Multiple Sclerosis Relapse (Nervous system disorders) | 1 | 0 | 2 | 1 — Treatment emergent = onset date is on or after the date of first dosing with IMP, and the onset date does not occur after the date of the Week 20 visit. Non-treatment emergent = onset date is after the date of the Week 20 visit.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intradermal Injection - Treatment Emergent (N=21) | Subcutaneous Injection - Treatment Emergent (N=22) | Intradermal Injection - Non Treatment Emergent (N=21) | Subcutaneous Injection - Non Treatment Emergent (N=22)
Injection Site Reactions (General disorders) | 12 | 7 | 0 | 0 — Treatment Emergent Adverse Event of mild to moderate intensity.
Nasopharyngitis (Infections and infestations) | 3 | 1 | 1 | 1 — Nasopharyngitis of mild to moderate intensity was experienced by 3 patients at the 800 μg dose level only (weeks 14 and 16).
Respiratory Tract Infection (Infections and infestations) | 2 | 0 | 1 | 0 — Emergent Adverse Events of moderate intensity.
Headache (Nervous system disorders) | 3 | 3 | 1 | 0 — Adverse Events of mild to moderate intensity.
Multiple sclerosis relapse (Nervous system disorders) | 2 | 3 | 4 | 4 — Adverse Events of moderate intensity. The number of MS relapses was not unexpected for this population.
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 — Adverse Events of mild intensity.
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 — Adverse Events of moderate intensity.
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 — Subject had a TEAE assessed as moderate in severity one week after the week 14 dose. This was located on the subject's back and arm whilst the injection was on the abdomen.
Anti-peptide Antibody response (Immune system disorders) | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If the Investigator drafts a publication, he/she agrees to send it to Apitope for review and comment before its submission to the journal. If Apitope considers that the proposed publication contains patentable material or information which should be protected as valuable confidential information, Apitope reserves the right to delay submission to the journal until patent applications have been filed and/or require the deletion of the confidential information from the proposed publication.